CLINICAL TRIAL: NCT05927987
Title: Feasibility and Acceptability of Problem Management Plus (PM+) for Prisoners in the Netherlands - a Pilot Randomised Controlled Trial
Brief Title: Feasibility and Acceptability of Problem Management Plus (PM+) for Prisoners in the Netherlands - a Pilot RCT
Acronym: PROSPER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: Netherlands Institute for the Study of Crime and Law Enforcement (NSCR) (Unknown)
Responsible Party: Principal Investigator, Mathilde van Oudenaren, PhD-student, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROSPER
Record Dates: First submitted 2023-06-13; First posted 2023-07-03 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Anxiety Disorders; Psychological Distress; Depressive Disorder
Keywords: Pilot Randomised Controlled Trial; Pilot RCT; Prisoner; Remand Prisoner; Remand custody; Prison; Dutch prison; Dutch prisons; PM+; Problem Management Plus; WHO intervention; Psychological Distress; Anxiety Disorder; Depressive disorder; Common Mental Health problems; Common Mental Health disorders
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: The RCT is a parallel-group, two-arm trial with a 1:1 allocation ratio. Participants are imprisoned adults in Dutch remand prisons with elevated levels of psychological distress (K10 > 15). Participants will be stratified by gender. A total of 60 participants will be included.
Who Masked: Outcomes Assessor
Masking Description: The participants will know to which group they are to be allocated. The PM+ supervisors, PM+ helpers, and two principal researchers will know which participants are randomised in a specific group. Involved research assistants (the outcome assessors) and the two other involved researchers will not know.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Problem Management Plus and care-as-usual (Experimental): The five sessions of PM+ will be delivered by trained master students in clinical psychology on an individual basis. Care-as-usual will not be withheld.
  Interventions: Behavioral: Problem Management Plus (PM+)
- Care-as-usual (No Intervention): Care-as-usual includes all social, health, and mental health services already available for individuals detained in Dutch prisons.

INTERVENTIONS:
Behavioral: Problem Management Plus (PM+) — Problem Management Plus (PM+) is a brief, psychological intervention program based on cognitive behavioural therapy (CBT) techniques that are empirically supported and formally recommended by the WHO (Dua et al., 2011; Tol et al., 2013). The full protocol was developed by the WHO and the University of New South Wales, Australia. The manual involves the following empirically supported elements: problem-solving, stress management, behavioural activation, and accessing social support. PM+ has three core features. It is brief (five sessions given in five weeks), delivered by paraprofessionals (PM+ helpers) and transdiagnostic. The PM+ helpers will be supervised by mental health care specialists.
  Arms: Problem Management Plus and care-as-usual

SUMMARY:
The goal of this pilot randomised controlled trial is to evaluate the feasibility and acceptability of the - specifically to the prison context adapted - World Health Organization's Problem Management Plus (PM+) intervention for individuals detained in Dutch remand prisons. The main question[s] it aims to answer are:

* To what extent is the contextually adapted PM+ intervention feasible and acceptable for individuals detained in Dutch remand prisons?
* To what extent are there preliminary indications of pre to post-effects of the PM+ intervention on, for example, anxiety and depression symptoms?

Researchers will compare two groups to answer these questions. Participants will either receive the PM+ intervention and Care-as-Usual or only Care-as-Usual.

DETAILED DESCRIPTION:
Rationale: Each year between 20 and 30 thousand individuals are newly incarcerated in Dutch prisons. Common mental disorders, such as depression and anxiety, are overrepresented in prison populations. As such, mental health problems are an important target for intervention, since they have been found to be associated with re-offending. The prison period may provide opportunities for addressing mental health problems, but there may be important obstacles and barriers to the actual delivery of interventions, such as a lack of mental health care specialists in prisons due to staff shortages.

Within the PROSPER study, we will evaluate the feasibility and acceptability of implementing the brief, scalable Problem Management Plus (PM+) intervention in Dutch prisons. The PM+ intervention is designed to address common mental health problems, is delivered by trained non-specialists, and will be specifically adapted for the prison setting.

Objective: The primary objective of the PROSPER study is to evaluate the feasibility and acceptability of PM+ adapted for individuals imprisoned in Dutch prisons.

Study design: This study entails a single-blind pilot randomised controlled trial (RCT) (Study Phase 2) and a qualitative study to evaluate the process following the pilot RCT (Study Phase 3).

Study population: Study Phase 2 - Dutch-speaking adults (18 years or older; N=60) who at the time of inclusion are enclosed in a Dutch remand prison and have a remaining sentence length of at least 15 weeks and who report an elevated level of psychological distress (K10 >15). Study Phase 3 - Participants (N= 20) will be from different stakeholder groups: the RCT participants, PM+ helpers, PM+ supervisors/trainers, and professionals. If permitted by RCT participants, family members, and friends are also invited.

Intervention (if applicable): Treatment group (n=30) - Participants in the treatment group will receive care-as-usual (CAU) and five sessions of PM+. PM+ is a brief, evidence-based psychological intervention and will be delivered by trained master students in clinical psychology and supervised by mental health care specialists. Control group (n=30) - This group will receive CAU only.

Main study parameters/endpoints: Main parameters are 1) PM+ fidelity, 2) perceptions about PM+ from stakeholders, 3) indicators of intervention delivery, 4) retention rate PM+ sessions, and 5) recruitment and consent rates. The secondary study parameter will be 1) symptoms of depression and anxiety (PHQ9 and GAD-7), 2) self-identified problems (PSYCHLOPS), 3) daily functioning (WHOQOL-BREF) and 4) symptoms of trauma (PCL-5) and suicidality vulnerability (SCOPE-2).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Study Phase 2 - participants enrolled in the treatment group will receive five sixty-minute PM+ sessions. If participants give permission, the sessions will be audiotaped for monitoring purposes. Additionally, all participants will be invited for a total of four assessments (one screening, one baseline assessment, and two post-intervention assessments). The post- intervention assessments will take place one week and three months after the last PM+ session. These assessments, all together, will take approximately 2 hours and 40 minutes. Study Phase 3 - Five stakeholder groups will be invited for individual interviews to evaluate the intervention and process. Each interview will take approximately 1 to 1,5 hours.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or above;
* Imprisoned in a Dutch prison;
* Held on remand;
* Dutch-speaking;
* Elevated levels of psychological distress (K10 >15);

Exclusion Criteria:

* Enclosed in a penitentiary psychiatric centre;
* Presents a potential security risk to the research team (PM+ helper and/or research team)
* Acute medical condition;
* Imminent suicide risk or expressed acute needs/protection risks (e.g., someone who expresses that they are at acute risk of being assaulted or killed);
* Severe mental disorder (psychotic disorders, substance dependence) ;
* Severe cognitive impairment (e.g., severe intellectual disability or dementia);
* Currently enrolled in a specialised psychological treatment program (e.g., EMDR, CBT);
* Less than two months on a stable dose of psychotropic medication (if applicable).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of PM+ | Outcomes are gathered throughout the study: during (factor 1) and after the trial finished (factors 2, 3, 4 and 5). We estimate inclusion will take about 9 months. Thus these factors will likely be gathered over a time frame of about one year.
  Factors relevant to the study of this outcome are:
  1. PM+ fidelity;
  2. The perceptions about PM+ from RCT participants, helpers, supervisors, trainers, professionals, and family members & friends of RCT participants;
  3. Indicators of intervention delivery, such as implementation process, adaptation, and dose.
  4. Retention rate PM+ sessions; and
  5. Recruitment and the consent rates.

SECONDARY OUTCOMES:
Preliminary indications of pre to post-effects on symptoms of depression and anxiety | Measured at baseline (week 0), week 8 and 13 weeks after baseline.
  Measured by Patient Health Questionnaire - 9 (PHQ9, depression) and Generalized Anxiety Disorder-7 (GAD-7, anxiety). A higher score on the PHQ9 (range = 1 - 27) means a greater severity of depressive symptoms. A higher score on the GAD-7 (range = 0 - 21) means a greater severity of anxiety symptoms.
Preliminary indications of pre to post-effects on self-identified problems | Measured at baseline (week 0), week 8 and 13 weeks after baseline.
  Measured by Psychological Outcome Profiles (PSYCHLOPS, self-identified problems). A higher score on the PSYCHLOPS (range = 0 - 20) means a greater severity of self-identified problems.
Preliminary indications of pre to post-effects on quality of life | Measured at baseline (week 0), week 8 and 13 weeks after baseline.
  Measured by World Health Organization Quality of Life Scale - brief (WHOQOL-BREF, quality of life). The score range differs per domain, but a higher score on every domain means a higher perceived quality of life. Domain I: 7 - 35. Domain II: 6 - 30. Domain III: 3 - 15. Domain IV: 8 - 40. Facet Overall Quality of Life and Health 2-10.
Preliminary indications of pre to post-effects on trauma | Measured at baseline (week 0), week 8 and 13 weeks after baseline.
  Measured by Post Traumatic Stress Disorder Checklist DSM5 (PCL-5, PTSD symptoms). A higher score on the PCL-5 (range = 0 - 80) means a greater severity of PTSD symptoms.
Preliminary indications of pre to post-effects on suicidal vulnerability | Measured at baseline (week 0), week 8 and 13 weeks after baseline.
  Measured by Suicide Concerns for Offenders in Prison Environment - 2 (SCOPE-2, suicidal vulnerability). A higher score on the SCOPE-2 (range = 19 - 76) means a greater vulnerability for suicide and non-fatal self-harm behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Marit EM Sijbrandij, PhD, Principal Investigator — Full professor - Vrije Universiteit Amsterdam
Locations (1):
- Vrije Universiteit Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dua T, Barbui C, Clark N, Fleischmann A, Poznyak V, van Ommeren M, Yasamy MT, Ayuso-Mateos JL, Birbeck GL, Drummond C, Freeman M, Giannakopoulos P, Levav I, Obot IS, Omigbodun O, Patel V, Phillips M, Prince M, Rahimi-Movaghar A, Rahman A, Sander JW, Saunders JB, Servili C, Rangaswamy T, Unutzer J, Ventevogel P, Vijayakumar L, Thornicroft G, Saxena S. Evidence-based guidelines for mental, neurological, and substance use disorders in low- and middle-income countries: summary of WHO recommendations. PLoS Med. 2011 Nov;8(11):e1001122. doi: 10.1371/journal.pmed.1001122. Epub 2011 Nov 15. PMID 22110406
- [Background] Tol WA, Barbui C, van Ommeren M. Management of acute stress, PTSD, and bereavement: WHO recommendations. JAMA. 2013 Aug 7;310(5):477-8. doi: 10.1001/jama.2013.166723. No abstract available. PMID 23925613
- [Background] de Graaff AM, Cuijpers P, Twisk JWR, Kieft B, Hunaidy S, Elsawy M, Gorgis N, Bouman TK, Lommen MJJ, Acarturk C, Bryant R, Burchert S, Dawson KS, Fuhr DC, Hansen P, Jordans M, Knaevelsrud C, McDaid D, Morina N, Moergeli H, Park AL, Roberts B, Ventevogel P, Wiedemann N, Woodward A, Sijbrandij M; STRENGTHS Consortium; STRENGTHS consortium. Peer-provided psychological intervention for Syrian refugees: results of a randomised controlled trial on the effectiveness of Problem Management Plus. BMJ Ment Health. 2023 Feb;26(1):e300637. doi: 10.1136/bmjment-2022-300637. Epub 2023 Feb 8. PMID 36789918
- [Background] Rahman A, Hamdani SU, Awan NR, Bryant RA, Dawson KS, Khan MF, Azeemi MM, Akhtar P, Nazir H, Chiumento A, Sijbrandij M, Wang D, Farooq S, van Ommeren M. Effect of a Multicomponent Behavioral Intervention in Adults Impaired by Psychological Distress in a Conflict-Affected Area of Pakistan: A Randomized Clinical Trial. JAMA. 2016 Dec 27;316(24):2609-2617. doi: 10.1001/jama.2016.17165. PMID 27837602
- [Derived] van Oudenaren MJF, Witteveen AB, Dirkzwager AJE, Sijbrandij M. Acceptability and feasibility of Problem Management Plus to address mental health problems among remand prisoners in the Netherlands: a pilot randomised controlled trial protocol. Health Justice. 2025 May 13;13(1):31. doi: 10.1186/s40352-025-00341-9. PMID 40358872
- See also: Individual Problem Management Plus manual — https://www.who.int/publications/i/item/WHO-MSD-MER-18.5